CLINICAL TRIAL: NCT04759794
Title: Clinical Validation of an Immunocytochemistry Method Using Antibody of Methionyl-tRNA Synthetase (MARS1) in the Bile Duct Cancer Cell; Multicenter Study
Brief Title: Clinical Validation of an Immunocytochemistry Method Using MARS1
Acronym: MARS1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Sung III Jang, Associate professor, Gangnam Severance Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3-2020-0514
Record Dates: First submitted 2021-02-15; First posted 2021-02-18 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Bile Duct Obstruction, Extrahepatic
Keywords: bile duct obstruction, extrahepatic; cytology; aminoacyl-tRNA synthetases
MeSH Terms: conditions — Cholestasis, Extrahepatic

STUDY DESIGN:
Intervention Model Description: The conventional staining method and new staining method will be performed in cytology specimens obtained from the same patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bile duct stenosis (Experimental): This arm includes patients with bile duct stenosis. Endobiliary brushing cytology specimens will be obtained with endoscopic retrograde cholangiopancreatography (ERCP) of patients with bile duct stenosis. Cytology staining will be performed in the cytology specimens.
  Interventions: Diagnostic Test: Cytology staining

INTERVENTIONS:
Diagnostic Test: Cytology staining — Two stainings will be performed in cytology specimens obtained from the same patient. The cytology specimen will be obtained through brushing cytology using endoscopic retrograde cholangiopancreatography
  1. conventional cytology staining method
  2. new cytology staining method using the antibody of aminoacyl-tRNA synthetases

SUMMARY:
The sensitivity of brushing cytology used to distinguish the cause of biliary strictures is low and clinical usefulness is not secured. The aim of this study was to validate the clinical usefulness of a new differential staining method for cytology which is difficult to differentiate by the conventional staining method using biliary cancer-related protein expressed only in bile duct cancer.

DETAILED DESCRIPTION:
Hypothesis: The statistical significance of new staining method using aminoacyl-tRNA synthetases (ARSs) group in normal bile duct cells and the bile duct cancer cells collected by endoscopic retrograde pancreaticoduodenoscopy (ERCP) will be compared to prove the usefulness of the new staining method.

Clinical study design: The bile duct cytology will be obtained by brushing cytology using ERCP in patients with biliary stenosis. The expression of ARSs in the brushing cytology will be evaluated by a new staining method and compare with the results of the conventional cytology staining method including Papanicolaou staining. Immunofluorescence or immunocytochemistry staining will be performed to differentiate the presence of the tumor. The sensitivity and specificity of the new staining method will be compared with the conventional staining method and its usefulness be confirmed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biliary cancer confirmed by imaging (CT, MRI, positron emission tomography)
* Patients with bile duct cancer diagnosed using brushing cytology by endoscopic retrograde pancreaticoduodenoscopy
* Patients who underwent surgical treatment with biliary cancer
* Patients with bile duct stenosis

Exclusion Criteria:

* Minors under the age of 19, vulnerable subjects such as illiteracy
* Necrotic specimens
* Samples with non-diagnostic cytology results and insufficient cells for further evaluation
* Samples classified as neoplastic (benign or other)
* Patient with cholangitis in the bile duct

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
The usefulness of new staining method | 1 year
  The sensitivity, specificity, positive predictive value, negative predictive value and accuracy of new staining method will be compared with th conventional Pap staining of brushing cytology specimens.

CONTACTS AND LOCATIONS:
Overall Officials: Sung Ill Jang, MD, PhD, Study Chair — Institutional Review Board, Gangnam Severance Hospital Yonsei University College of Medicine
Locations (5):
- South Korea (5):
  - CHA Bundang Medical Center, Seongnam, Bundang-gu
  - Gangnam Severance Hospital, Seoul, Gangnam-gu
  - In Ha University Hospital, Incheon, Jung-gu
  - Soon Chun Hyang University Hospital, Cheonan, Cheonan, Namdong-gu
  - Pusan National University Hospital, Busan, Seo-gu

IPD SHARING:
Plan to Share IPD: Yes
We plan to share the following individual participant data with other researchers during the study period.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 1 year
Access Criteria: * Primary investigator
  * Sub primary investigator